CLINICAL TRIAL: NCT06723951
Title: Validation of the Quality of Life Assessment in Spina Bifida for Children and Adolescents in Dutch
Brief Title: QUALAS Validation in Dutch
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Lisette 't Hoen, Principal Investigator, Erasmus Medical Center
Other Study IDs: EMCSophia2
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Spina Bifida
MeSH Terms: conditions — Spinal Dysraphism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Children with spina bifida: • Male or female aged 8 -12 years with spina bifida
  Interventions: Other: QUALAS survey
- Control group children: • Male or females aged 8 -12 years without spina bifida
  Interventions: Other: QUALAS survey
- Teenagers with spina bifida: • Males or female aged 13 - 17 years with spina bifida
  Interventions: Other: QUALAS survey
- Control group teenagers: • Males or females aged 13 - 17 years without spina bifida
  Interventions: Other: QUALAS survey
- Adults with spina bifida: Adults with spina bifida
  Interventions: Other: QUALAS survey
- Control group adults: Adults without spina bifida
  Interventions: Other: QUALAS survey

INTERVENTIONS:
Other: QUALAS survey — Participants will be asked to complete the surveys at one (controls) and two (patients) timepoints.
  Other Names: KIDSCREEN survey for children and teenagers; World Health Organization Quality of Life instrument (WHOQOL-BREF) and (International Consultation on Incontinence Questionnaire) ICIQ for adults

SUMMARY:
Rationale Patients with spina bifida often experience a decreased quality of life compared to patients without spina bifida. The Quality of Life Assessment for Spina Bifida (QUALAS) is a validated questionnaire to assess the quality of life in children, teenagers and adults with spina bifida, accounting for specific factors, such as bladder and bowel dysfunction. This questionnaire enables us to assess the current spina bifida related quality of life and identify if bladder and bowel dysfunction is of influence.

Objective(s) To validate the Quality of Life Assessment for Spina Bifida in Children, Teenagers and Adults in Dutch.

Study type A multicenter prospective validation cohort study.

Study population Children aged 8 - 17 years and adults who are diagnosed with spina bifida. As a control group children aged 8 - 17 years and adults without spina bifida will be approached at the Ear-Nose-Throat (ENT) and paediatric clinics.

Methods The main study parameter is the validation of the Dutch version of the questionnaire. Patients with spina bifida are asked to fill out the QUALAS at two time-points. They are also asked to fill out an extra questionnaire at two time-points, in order to validate the QUALAS. Children and adults in the control groups are asked to fill out the two questionnaires only once.

Burden and risks No (extra) outpatient visit is required. The questions in the questionnaires are similar to the medical history during an outpatient visit. The burden is therefore minimal for these patients. Participation in this study will not influence patient treatment.

Recruitment and consent Parents of children and children and adults who meet the inclusion criteria and none of the exclusion criteria will be informed orally about this study by their treating urologist during a regular visit. A patient information and consent form will be handed over to the parents and children over eight years of age and adults. Parents of children and children and adults at the ENT clinic will be approached by the local urologist for participation for this study. If they are willing to participate they will be asked to sign informed consent and fill out the questionnaire.

DETAILED DESCRIPTION:
Introduction and rationale Patients with spina bifida often face challenges in different areas. It is common to have a dedicated team of medical specialists for yearly follow-up. This team includes paediatricians, neurosurgeons, orthopaedics, urologists and rehabilitation specialists. Patients with spina bifida may experience symptoms in each of these areas which will have an impact of these patient's quality of life. From the urologist perspective urinary incontinence and faecal incontinence have a high impact on quality of life.

Questionnaires to evaluate quality of life in patients with spina bifida do not incorporate these specific symptoms. The QUAlity of Life Assessment in Spina bifida in Children (QUALAS-C), QUAlity of Life Assessment in Spina bifida in Teenagers (QUALAS-T) and The QUAlity of Life Assessment in Spina bifida in Adults (QUALAS-A) have been developed to take these symptoms into account when assessing quality of life. These questionnaires are validated in the United States. For children aged 8-12 years the QUALAS-C version is available. For children between 13-17 years of age the QUALAS-T version is available. For adults the QUALAS-A version is available.

Currently, no versions of the QUALAS-C, QUALAS-T, QUALAS-A questionnaires are available in Dutch.

With the QUALAS-C, QUALAS-T and QUALAS-A the investigators will be able to assess spina bifida related quality of life and monitor the development over time. This will enable clinicians to offer improved standardized care.

Objective(s) The aim of this study is to validate the QUALAS questionnaire for children, teenagers and adults in Dutch.

Methods This is a multicenter prospective cohort validation study of the QUALAS questionnaire. This is a spina bifida related quality of life questionnaire. The investigators will validate the QUALAS using the validated KIDSCREEN-27 for children 8-17 years of age and the World Health Organization Quality of Life instrument (WHOQOL-BREF) and (International Consultation on Incontinence Questionnaire) ICIQ for adults questionnaires to determine spina bifida related quality of life in a standardized manner.

All patients are subject to treatment at the department of Paediatric Urology in Erasmus MC-Sophia or University Medical Center Groningen. Participation in this study will not interfere with their treatment.

For this study two different phases are distinguished:

* Phase 1: The QUALAS will be translated following a standardized translation process. This includes three forward translations by Dutch native speakers, one backward translation by a English native speaker and face-to-face testing in the target population.
* Phase 2: Children of 8 years and older and adults are asked to fill out the questionnaires, QUALAS and KIDSCREEN for children 8-17 years of age and the WHOQOL-BREF and ICIQ for adults, and repeat filling out the QUALAS questionnaire one week later. The team asks all parents to fill out the questionnaire in order to secure a constant answer during the study. Children of 8 years and older and adults in the control group are asked to fill out the QUALAS and KIDSCREEN-27 for children 8-17 years of age and the WHOQOL-BREF and ICIQ for adults. Internal consistency, criterion validity, construct validity an reproducibility will be determined.

ELIGIBILITY:
Inclusion Criteria:

Patient group:

* Male or female patients aged 8 -12 years (QUALAS-C)
* Male or female patients aged 13 - 17 years (QUALAS-T)
* Adult patients (QUALAS-A)
* Has spina bifida
* Adult or child and at least one parent fluent in the Dutch language
* Signed informed consent

Control group:

* Male or female children aged 8 -12 years (QUALAS-C)
* Male or female adolescents aged 13 - 17 years (QUALAS-T)
* Adults (QUALAS-A)
* Has no spina bifida
* Adult or child and at least one parent fluent in the Dutch language
* Signed informed consent

Exclusion Criteria:

* Has a neurogenic disease other than spina bifida
* Has had surgery in the last month

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents of children and children and adults with spina bifida that are patients at the Urology department of the two hospitals will be approached to participate.
  This questionnaire quantifies the quality of life in patients with spina bifida, with a special interest in bladder and bowel dysfunction.
  A group of children and adults without spina bifida will function as a control group. These children and adults will be approached at the ENT and paediatric clinics.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-09 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Internal consistency of QUALAS | 3 months
  Internal consistency is the main study endpoint. This will be calculated with Cronbach's alpha. Values between 0.70 and 0.95 reflect good consistency.
  QUALAS questionnaire:
  Scores range from 0-100 with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Reproducibility | 2 weeks
  Reproducibility will be determined to assess the ability to reproduce similar answers during the retest period. This will be calculated using Intraclass Correlation Coefficient (ICC), where ICC scores over 0.7 are acceptable. The limits of agreement (LOA), which is calculated by mean change in scores ± 1.96 SD are determined as well.
Content validity | 3 months
  Content validity is subjectively determined by examining whether the questionnaire is measuring the quality of life related to spina bifida.
Construct validity | 3 months
  Construct validity is determined by testing the following hypotheses:
  * The control group will have higher scores in the QUALAS than patients with spina bifida.
  * Patients who score higher in the KIDSCREEN-27 or WHOQOL-BREF/ICIQ will have higher scores in the QUALAS.
  The KIDSCREEN-27: Each item is scored on a 5-point Likert scale ranging from 1 meaning "not at all" to 5 meaning "very much". Certain items (1, 9, 10 and 11) were reversed when scoring the questionnaire. Reverse scoring means that the numerical scoring scale runs in the opposite direction. The total KIDSCREEN score was calculated by summing up all the responses. Higher scores of KIDSCREEN indicated better QoL and social support.
  The WHOQOL-BREF questionnaire: 26 items are scored on a 5-point Likert scale. Scores range from 0-100 with higher scores indicating better quality of life
  The ICIQ questionnaire: 3 items are scored with a total sum range of 0-21, higher score indicate worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Lisette 't Hoen, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (2):
- Netherlands (2):
  - UMCG, Groningen
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT06723951/Prot_000.pdf